CLINICAL TRIAL: NCT07141797
Title: Impact of General Anesthesia in Childhood on Cognitive Processes
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00110-83
Record Dates: First submitted 2025-07-02; First posted 2025-08-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Neurodevelopmental Disorders; Child Behavior Disorders
Keywords: general anesthesia; children; developing brain; executive functions; cognitive assessment
MeSH Terms: conditions — Neurodevelopmental Disorders; Child Behavior Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anesthesia group: Children aged 9 or 10 at the time of the study, who were exposed to a single general anesthesia for a functional surgery during childhood before the age of 4.
  Interventions: Other: Executive functions assessment
- Control group: Children aged 9 or 10 at the time of the study, who were not exposed to general anesthesia for surgery during childhood.
  Interventions: Other: Executive functions assessment

INTERVENTIONS:
Other: Executive functions assessment — Inhibition: Emotional (hot) and logical (cold) inhibition using Emotional and Classic Stroop tests. Participants identify the color of words or emotion in photos while inhibiting automatic responses. Inhibition scores are based on the difference in response times between congruent and interference conditions.
  Working Memory: Participants recall a sequence of points on a grid, first in the original order, then in reverse. The working memory score is the difference between the two tasks.
  Cognitive Flexibility: A task requiring alternation between identifying numbers as greater/less than 5 or even/odd based on color cues. Flexibility is scored by comparing response times for alternating and non-alternating tasks.
  Visuospatial abilities are assessed with a global-local task. Raven's Progressive Matrices will assess general intelligence, and socio-economic data will be collected.

SUMMARY:
This study aims to evaluate the potential long-term cognitive effects of general anesthesia administered before the age of 4. Specifically, it investigates executive functions-including inhibition, working memory, and cognitive flexibility-in children aged 9 to 10 years. A secondary objective assesses visuo-spatial attention.

Participants will be divided into two groups: (1) children exposed to a single general anesthesia for functional surgery before age 4, and (2) a control group with no such exposure. Cognitive performance will be assessed through computerized tasks with time constraints, conducted in a school setting. The study is designed to compare these groups prospectively in order to determine whether early exposure to general anesthesia is associated with differences in cognitive functioning at school age.

DETAILED DESCRIPTION:
This study investigates the long-term cognitive effects of early exposure to general anesthesia in children. Specifically, it focuses on evaluating executive functions-namely inhibition, working memory, and cognitive flexibility-in children aged 9-10 years who underwent functional surgery with general anesthesia before age 4. A secondary objective includes assessing visuo-spatial attention and general intelligence.

Executive functions will be measured using standardized, computerized tasks. Inhibition will be assessed through both an emotional Stroop (hot inhibition) and a classic Stroop task (cold inhibition). Working memory will be evaluated using a spatial sequence recall task on a grid, in both forward and reverse order. Flexibility will be measured through an adapted version of the computerized Trail Making Test, requiring rule-switching between tasks based on stimulus color.

Visuo-spatial abilities will be assessed using a global-local task involving hierarchical visual stimuli, allowing for evaluation of attention to detail versus overall structure. General intelligence will be measured using Raven's Progressive Matrices.

Participants will be recruited from selected elementary schools in partnership with local educational authorities. Eligible children will be grouped based on prior exposure to general anesthesia, matched on age, sex, and socio-economic status. Testing will occur in school settings during class time under controlled, blinded conditions. Data will be anonymized and processed in accordance with GDPR standards. Statistical analyses will include MANOVA and linear models to assess group differences.

ELIGIBILITY:
Inclusion Criteria:

Children aged 9-10 years Mainstream class (non-specialized) Requirement for information on the right to object Requirement for affiliation with social security French-speaking

Exclusion Criteria:

Criteria for "Parents" Parental refusal Twins Exposure to general anesthesia during pregnancy, including cesarean section under general anesthesia

Pregnancy-related pathology:

* Pregnancy-induced hypertension
* Preeclampsia
* Gestational diabetes
* Threat of preterm labor
* Depressive syndrome

Chronic treatment during pregnancy:

* Pregnancy-induced hypertension: antihypertensive treatment (beta-blockers, calcium channel blockers)
* Preeclampsia: antihypertensive treatment (beta-blockers, calcium channel blockers), magnesium sulfate
* Gestational diabetes: dietary regimen, insulin
* Threat of preterm labor: prenatal corticosteroid therapy, magnesium sulfate
* Depressive syndrome: antidepressant psychotropic treatment Smoking during pregnancy, alcohol consumption during pregnancy, drug use during pregnancy Criteria for "Children" Child refusal to participate in the study Premature birth (i.e., before 37 weeks of gestation) Evolving or chronic psychiatric pathology, whether or not requiring chronic treatment Evolving or chronic neurological or neuromuscular pathology Genetic pathology Any chronic pathology requiring specialized follow-up and/or treatment (doctor, psychologist, speech therapist) Specialized neuro-pediatric or pediatric psychiatric follow-up, or follow-up with a psychologist or speech therapist during childhood Neuro-visual disorders (excluding normal vision with correction) Hearing disorders, whether or not using hearing aids Chronic otorhinolaryngological pathology, including sleep apnea syndrome, with or without apparatus Developmental disorders: ADHD, autism, or other, whether or not requiring chronic treatment Pediatric intensive care hospitalization Conventional hospitalization for more than 1 week during childhood Child who underwent multiple general anesthesias before the age of 4

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 9-10 years, attending school, who have either been exposed or not exposed to general anesthesia for a functional surgery before the age of 4.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Inhibition/ working memory/ flexibility | Day 1 (single school testing session). The assessment of all judgment criteria is conducted during a 30-minute timed testing session on a computer, with the child present.
  Cold Inhibition: Measured by the Stroop task (color-word interference). Unit: reaction time difference (ms).
  Hot Inhibition: Measured by the emotional Stroop (faces and emotional words). Unit: reaction time difference (ms).
  Working Memory: Assessed via forward and backward spatial recall on a grid. Unit: number of correct sequences.
  Cognitive Flexibility: Measured by a rule-switching task (digit color cues: magnitude vs. parity). Flexibility is the RT difference between switch and control tasks. Unit: reaction time difference (ms).

SECONDARY OUTCOMES:
Visuo-spatial abilities/ measure of general intelligence | Day 1 (single school testing session). The assessment of all judgment criteria is conducted during a 30-minute timed testing session on a computer, with the child present.
  Visuo-spatial abilities will be assessed using a global-local task, where participants identify shapes (square or circle) at either the global or local level, based on hierarchical stimuli. This evaluates attentional processing of visual details vs. overall structure. A general intelligence test will also be administered to ensure group equivalence.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Caen Normandie, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided